CLINICAL TRIAL: NCT01256047
Title: Effects of Preoperative Immunonutrition on Infectious Complication and Th1/Th2 Differentiation in Patients Undergoing Hepatectomy
Brief Title: Effects of Preoperative Immunonutrition in Patients Undergoing Hepatectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chiba University (Other)
Responsible Party: Principal Investigator, Katsunori Furukawa, MD, PhD, Chiba University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: furukawa2009-2
Record Dates: First submitted 2010-12-07; First posted 2010-12-08 (Estimated); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Bile Duct Cancer
Keywords: immunonutrition; hepatectomy; Th1; Th2
MeSH Terms: conditions — Bile Duct Neoplasms | interventions — Long-Term Synaptic Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- group A (Active Comparator): preoperative immunonutrition
  Interventions: Dietary Supplement: Oral IMPACT
- group B (No Intervention): ordinary diet

INTERVENTIONS:
Dietary Supplement: Oral IMPACT — oral supplement for 5 days(1L/day) before surgery of a formula enriched with arginine, omega-3 fatty acids, and RNA
  Other Names: Oral IMPACT; Ajinomoto Pharma Co., Ltd, Tokyo, Japan
  Arms: group A

SUMMARY:
The purpose of this study is to determine whether preoperative immunonutrition is effective on infectious complication and Th1/Th2 differentiation in patients with major hepatectomy.

DETAILED DESCRIPTION:
The investigators reported that preoperative immunonutrition improve the incidence of postoperative infectious complication in patients after hepatectomy, and modulation of Th1/Th2 differentiation may play important roles in this effect.

Object of this study is to investigate the effects of preoperative immunonutrition on incidence of postoperative infectious complication, and Th1/Th2 balance after hepatectomy.

ELIGIBILITY:
Inclusion Criteria:

* hepatectomy

Exclusion Criteria:

* age younger than 18 years
* ongoing infection
* gastrointestinal obstruction
* respiratory dysfunction
* cardiac dysfunction
* hepatic dysfunction
* renal failure
* history of recent immunosuppressive or immunological disease
* preoperative evidence of widespread metastatic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-05; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
postoperative infectious complication | 30 days

SECONDARY OUTCOMES:
plasma IL-6, CRP, Th1/Th2 balance | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Katsunori Furukawa, MD, Study Director — Chiba University
Locations (1):
- Chiba University, Chiba, Japan

REFERENCES:
- [Derived] Uno H, Furukawa K, Suzuki D, Shimizu H, Ohtsuka M, Kato A, Yoshitomi H, Miyazaki M. Immunonutrition suppresses acute inflammatory responses through modulation of resolvin E1 in patients undergoing major hepatobiliary resection. Surgery. 2016 Jul;160(1):228-236. doi: 10.1016/j.surg.2016.01.019. Epub 2016 Mar 8. PMID 26965712